CLINICAL TRIAL: NCT02035852
Title: High Resolution Magnetic Resonance Imaging in Patients With Brain Tumors
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: STU 062010-160; 1R01CA154843-01A1 (NIH)
Record Dates: First submitted 2012-06-12; First posted 2014-01-14 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-11

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adult Gilomas
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — 3T MRI vs. 7T MRI

SUMMARY:
The study will compare two different size MRI's of a brain tumor.

DETAILED DESCRIPTION:
The study is designed to directly compare the MR images of a brain tumor obtained on the 3T and then 7T MRI in approximately 150 patients followed serially with MR imaging to evaluate for tumor progression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older
* Patient must meet at least one of the four following criteria regarding brain tumor diagnosis:
* Histological diagnosis of a brain tumor
* Histological diagnosis of systemic cancer and brain MR imaging suggestive of metastatic disease to the brain
* Pre-operative brain MR imaging suggestive of a brain tumor
* Radiographic diagnosis of brain tumor in an inoperable location (e.g., brainstem)
* Patient able and willing to provide informed consent
* Karnofsky Performance status > 70%
* Life expectancy greater than 3 months
* Negative serum or urine pregnancy test or child bearing potential terminated by surgery, radiation, menopause or current use of two approved methods of birth control
* Patients who are excluded from 7T MR imaging because of titanium implants that are not yet established to be safe at 7T remain eligible for the imaging at 3T * Spanish speaking participants will be enrolled for this study

Exclusion Criteria:

* Body weight >137 Kg (300 lbs)
* Patient unable to provide informed consent
* Karnofsky Performance status < 70%
* Patients who are claustrophobic or have other contraindications to MRI, such as implanted pacemaker device vascular clips, surgical clips, prosthetic valves, pacemakers, otologic implants
* NYHA class III and IV congestive heart failure
* Psychiatric or addictive disorders that preclude obtaining informed consent
* Unstable angina
* Sexually active patients of childbearing potential not using a reliable contraceptive method
* Pregnant or lactating women
* Women of childbearing potential who refuse a pregnancy test (performed during screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the Simmons Cancer Center at UTSW
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2009-08-28 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Benefit of 7T MR imaging | Baseline and 6 month intervals after baseline
  1. To determine the benefit of 7T MR imaging in brain tumor patients with regard to the improvement in resolution, as measured by the area of T2 FLAIR signal abnormality and the ability to detect abnormalities in vascular integrity. The benefit will be determined at a single time point as well as longitudinally for each patient at 6 month intervals.

SECONDARY OUTCOMES:
Vascular Integrity | Every 6 months, up to 12 months.
  To determine if changes in vascular integrity at 7T can be correlated with tumor progression or transformation to high grade in patients with low grade gliomas.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Maher, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States